CLINICAL TRIAL: NCT07372755
Title: Feasibility and Usability of a Mobile App for Monitoring and Managing Functional Movement Disorders
Status: Not yet recruiting | Type: Observational
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Aditya Murgai, Assistant Professor, Western University, Canada
Other Study IDs: 128351
Record Dates: First submitted 2026-01-19; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Functional Movement Disorder
Keywords: functional movement disorder; mobile app
MeSH Terms: conditions — Conversion Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Functional Movement Disorder

SUMMARY:
People with FMD may experience symptoms such as tremor, jerks, spasms, or difficulty walking. These symptoms are not caused by damage to the brain or nerves. Instead, they happen because the brain is not sending or processing signals in the usual way. Symptoms can change from day to day, and stress, emotions, or certain situations may make them better or worse.

Right now, patients are often asked to remember how their symptoms have been since their last clinic visit or to write things down in a notebook. This can be hard to do and may not give an accurate picture of what is happening. Because of this, doctors and patients may miss important patterns or triggers, and it can be harder to know which coping strategies are helpful.

To improve this, our team has created a mobile app that allows people with FMD to easily record their symptoms, stress level, and mood, in real time. The app also includes simple self-help tools that may support symptom management. Before using this app more widely, we want to find out (1) whether patients can use it as intended and (2) whether they find it easy and helpful to use. This study will help us understand if the app is practical for use in an FMD clinic and how it could be improved.

DETAILED DESCRIPTION:
Functional movement disorders (FMD) can cause symptoms such as tremor, jerking, or walking difficulties. These symptoms are not due to structural damage in the brain or nerves but relate to how the brain is functioning. Symptoms often vary over time and may be affected by stress, emotions, and everyday situations, which can be hard to track accurately between clinic visits.

This study will evaluate the feasibility and usability of a mobile application designed to help people with FMD record symptom flares, stress levels, and possible triggers, and access simple self-help tools. The app also produces summary reports that can be reviewed during clinic visits.

Ten adults with FMD will use the app for six weeks. Participants on the first visit will be given brief training about the app. Follow-up visits will be every two weeks to review app summaries and address technical issues. At week 6, participants will complete a short usability questionnaire and a brief interview about their experience.

The study's main goal is to determine whether participants can and will use the app as intended and whether they find it acceptable and easy to use

We invite you to take part in a research study looking at a new mobile phone app designed for people with Functional Movement Disorders (FMD). Taking part is completely voluntary.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18
* Diagnosed with a functional movement disorder
* Own a smartphone
* Ability to read and understand English
* Ability to provide informed consent

Exclusion Criteria:

* Acute psychiatric crisis
* Limitations that make it impossible to use a smartphone app

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Functional Movement Disorder Clinic
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Can patients use the app as intended for 6 weeks? | 6 weeks
  Can patients use the app as intended for 6 weeks?
Acceptability and Usability | 6 weeks
  Do patients find the app acceptable and easy to use?

SECONDARY OUTCOMES:
Clinical Utility | 6 weeks
  Do app summaries feel clinically useful during visits?

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, London, Canada

IPD SHARING:
Plan to Share IPD: No
At this time, IPD will not be shared due to confidentiality concerns.